CLINICAL TRIAL: NCT07153289
Title: Response Features, Efficacy and Safety of CD318-targeted CAR-T Cell Therapy Against Pancreatic Cancer - ResCPa Study
Brief Title: CD318-targeted CAR-T Cell Therapy in Patients With Pancreatic Cancer (ResCPa)
Acronym: ResCPa
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: University Hospital Freiburg (Other); Technical University of Munich (Other); National Center for Tumor Diseases, Heidelberg (Other); Wuerzburg University Hospital (Other); Berlin Institute of Health (Other); Miltenyi Biotec B.V. & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-523195-23-00; 01KD2421A (Other Grant/Funding Number: Federal Ministry of Education and Research (BMBF))
Record Dates: First submitted 2025-08-08; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Carcinoma, Pancreatic Ductal; Pancreatic Neoplasms
Keywords: PDAC; Metastatic Pancreatic Cancer; Locally Advanced Pancreatic Cancer; CD318 CAR-T; CAR-T cell therapy
MeSH Terms: conditions — Carcinoma, Pancreatic Ductal; Pancreatic Neoplasms | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Intervention Model Description: Sequential single-group design: Phase I dose escalation (single infusion) followed by a Phase IIa expansion cohort at RP2D with dual dosing. Participants are not assigned in parallel to different regimens.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD318-CAR-T: Phase I dose escalation with Phase IIa expansion (dual dosing) (Experimental): Single experimental cohort receiving autologous CD318-targeted CAR-T cells after lymphodepletion. The study proceeds sequentially in two stages: (1) Phase I dose escalation using a Bayesian Optimal Interval (BOIN) design to determine the maximum tolerated dose (MTD) and/or recommended phase II dose (RP2D) with a single infusion; (2) Phase IIa expansion at the RP2D employing a predefined dual-dosing schedule (two infusions) to further evaluate safety and preliminary efficacy. Participants are not assigned in parallel to different regimens.
  Interventions: Biological: CD318-CAR-T cells

INTERVENTIONS:
Biological: CD318-CAR-T cells — Autologous T cells collected by leukapheresis, genetically modified using a GMP-manufactured lentiviral vector encoding a fully human CD318-specific chimeric antigen receptor (CAR), and expanded on the CliniMACS Prodigy system. After lymphodepleting chemotherapy (fludarabine/cyclophosphamide), participants receive (Phase I) a single CAR-T infusion per BOIN dose-escalation to determine MTD/RP2D; (Phase IIa) an expansion at RP2D with a predefined dual-dosing schedule (two infusions) separated by a protocol-defined interval.
  Other Names: ResCPa, CD318 CAR-T, CD318-CAR, CAR-T cell therapy

SUMMARY:
Pancreatic ductal adenocarcinoma (PDAC) is one of the most lethal cancers, with limited therapeutic options and a five-year survival rate below 10 % in advanced stages. Standard treatments, such as multi-agent chemotherapy, provide only marginal survival benefits and are often associated with significant toxicity. Novel approaches are urgently needed.

The ResCPa study is a first-in-human, multicenter, phase I/IIa investigator-initiated trial evaluating the safety, feasibility, and preliminary efficacy of autologous CD318-targeted chimeric antigen receptor (CAR) T-cell therapy in patients with metastatic or locally advanced PDAC that has progressed after standard-of-care treatment. CD318 (also known as CDCP1) is highly expressed in primary and metastatic PDAC tissue but rarely found in healthy tissues, making it a promising and potentially safe immunotherapy target. Preclinical studies have shown potent anti-tumor activity of CD318-CAR-T cells in vitro and in PDAC mouse models without target-specific toxicity.

Eligible patients will undergo tumor tissue screening for CD318 expression. Those meeting the criteria will proceed to leukapheresis for autologous T-cell collection. The CD318-CAR construct, optimized in preclinical work, will be introduced via a GMP-produced lentiviral vector, and CAR-T cells will be expanded using automated manufacturing (CliniMACS Prodigy). Following lymphodepleting chemotherapy, patients will receive CD318-CAR-T cells in a dose-escalation design to determine the recommended phase II dose, with the option of dual dosing.

The primary objectives are to assess safety, tolerability, and feasibility of manufacturing and delivering CD318-CAR-T cells. Secondary objectives include preliminary anti-tumor activity (objective response rate, progression-free survival, overall survival), CAR-T cell expansion and persistence, and immunological correlates of response or resistance. Patients will be followed for at least 12 months post-infusion, with extended safety follow-up per regulatory requirements.

In parallel, an extensive translational research program will investigate CAR-T cell phenotypes, tumor microenvironment changes, and mechanisms of treatment resistance using single-cell multi-omics, spatial proteomics and transcriptomics, organoid co-culture models, and microbiome profiling. Insights from these studies aim to guide optimization of next-generation CAR-T therapies for PDAC and other solid tumors.

This trial is conducted by a German academic-industrial consortium including the University Hospital Tübingen, Miltenyi Biotec, University Hospital Freiburg, Klinikum rechts der Isar (TUM), Berlin Institute of Health (BIH), and other partners. The study is supported by the German Federal Ministry of Education and Research (BMBF) within the "National Decade Against Cancer" initiative.

DETAILED DESCRIPTION:
Pancreatic ductal adenocarcinoma (PDAC) is one of the most lethal malignancies, with a steadily increasing incidence and a poor prognosis. Standard chemotherapy regimens such as FOLFIRINOX or gemcitabine plus nab paclitaxel provide only modest survival benefits and are often associated with substantial toxicity. PDAC is characterized by aggressive tumor biology, early metastasis, and marked resistance to conventional therapies, underscoring the need for novel strategies.

Chimeric antigen receptor (CAR) T cell therapy has transformed the treatment of hematologic malignancies but has yet to achieve similar success in solid tumors. Challenges include the lack of highly specific tumor antigens, poor trafficking and persistence of CAR T cells, immune evasion in the tumor microenvironment, and tumor antigen heterogeneity.

CD318, also known as CDCP1, is a promising target for PDAC immunotherapy. It is highly expressed in primary and metastatic PDAC tissues but shows minimal expression in healthy tissues. Preclinical studies have demonstrated that CD318 targeted CAR T cells can induce potent anti tumor activity in vitro and in PDAC mouse models without detectable target specific toxicity.

The ResCPa study is a first in human, multicenter, phase I/IIa investigator initiated clinical trial designed to evaluate the safety, feasibility, and preliminary efficacy of autologous CD318 targeted CAR T cells in patients with metastatic or locally advanced PDAC refractory to standard of care therapy. The study will also conduct an extensive translational research program to understand CAR T cell function and resistance mechanisms in solid tumors.

Eligible patients will be screened for CD318 expression in tumor tissue. Those meeting inclusion criteria will undergo leukapheresis for T cell collection. Autologous T cells will be genetically modified using a GMP manufactured lentiviral vector encoding the CD318 CAR and expanded using automated manufacturing on the CliniMACS Prodigy platform at the University Hospital Tuebingen GMP facility.

Following lymphodepleting chemotherapy, patients will receive CAR T cells in a dose escalation design using the Bayesian Optimal Interval method to determine the maximum tolerated dose or recommended phase II dose. Dose limiting toxicities will be closely monitored and predefined stopping rules applied. Both single and dual dosing regimens may be used.

Primary objectives are to assess the safety, tolerability, and feasibility of manufacturing and delivering CD318 CAR T cells. Secondary objectives are to evaluate preliminary antitumor activity, CAR T cell expansion and persistence, and immune correlates of response or resistance. Exploratory objectives include biomarker discovery, characterization of the tumor microenvironment, and microbiome analyses.

Translational research will include

* Immune monitoring by single cell multi omics profiling of CAR T cell products and longitudinal blood samples to evaluate phenotype, activation status, metabolic fitness, and exhaustion markers.
* Tumor microenvironment analyses using spatial proteomics, spatial transcriptomics, and imaging mass cytometry of tumor biopsies before and after treatment to assess immune infiltration, antigen expression, and stromal architecture.
* Patient derived organoid and xenograft models to study CAR T cytotoxicity, antigen recognition, and resistance mechanisms in vitro and in vivo.
* Microbiome profiling of stool and tumor samples using shotgun metagenomics and 16S rRNA sequencing to explore associations with response or resistance.
* Characterization of innate like T cell subsets such as gamma delta T cells, NKT cells, and MAIT cells within CAR T products and exploration of CD318 targeting in these populations.

The trial is coordinated by the University Hospital Tuebingen in collaboration with Miltenyi Biotec, University Hospital Freiburg, Klinikum rechts der Isar TUM, Max Delbrueck Center Berlin, and other partners. It is funded by the German Federal Ministry of Education and Research BMBF under the National Decade Against Cancer initiative. A Data Safety Monitoring Board will oversee patient safety, and a patient advisory board will be involved in study oversight and dissemination of results.

If successful, this trial could establish CD318 CAR T therapy as a new treatment option for PDAC and provide insights to optimize future CAR T approaches for solid tumors. Findings may also have relevance for other cancer types, accelerating the development and clinical application of advanced cellular immunotherapies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the time of informed consent
* Histologically confirmed PDAC (metastatic or locally advanced, unresectable)
* Measurable disease according to RECIST v1.1
* Disease progression during or after at least one prior line of systemic standard therapy for advanced PDAC
* CD318 expression in tumor tissue confirmed by central immunohistochemistry (IHC)
* ECOG performance status of 0 or 1
* Adequate bone marrow, renal, and hepatic function as defined in the protocol
* Life expectancy of at least 12 weeks
* Willingness and ability to comply with study procedures and follow-up
* Written informed consent obtained prior to any study-specific procedures-

Exclusion Criteria:

* Prior treatment with CAR T cells or other genetically modified cell therapies
* Active uncontrolled infection, including active hepatitis B or C infection or HIV infection
* Known symptomatic or untreated central nervous system (CNS) metastases
* Clinically significant cardiovascular disease, including recent myocardial infarction (within 6 months), unstable angina, or uncontrolled arrhythmia
* History of autoimmune disease requiring systemic immunosuppressive therapy
* Current or recent (within 4 weeks) participation in another interventional clinical trial
* Pregnant or breastfeeding women
* Any condition that, in the opinion of the investigator, would interfere with the patients ability to comply with study requirements or would compromise safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of dose-limiting toxicities (DLTs) and adverse events (AEs) after CD318-CAR-T cell infusion. | From CAR-T cell infusion through Day 28 after the last infusion in each subject.
  Assessment of safety and tolerability of autologous CD318-CAR-T cells by determining the incidence, severity, and relationship to treatment of DLTs and AEs, graded according to NCI CTCAE version 5.0.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 12 months after CAR-T cell infusion.
  Proportion of patients achieving complete or partial response as best overall response, assessed by RECIST v1.1 and/or iRECIST criteria.
Duration of response (DoR) | Up to 12 months after CAR-T cell infusion.
  Time from first documented response (complete or partial) to documented disease progression or death from any cause, whichever occurs first.
Progression-free survival (PFS) | Up to 12 months after CAR-T cell infusion.
  Time from CAR-T cell infusion to disease progression per RECIST v1.1/iRECIST or death from any cause.
Overall survival (OS) | Up to 12 months after CAR-T cell infusion, with potential long-term follow-up per protocol.
  Time from CAR-T cell infusion to death from any cause.
CAR-T cell expansion and persistence in peripheral blood | From infusion until Month 12 post-infusion.
  Quantification of CD318-CAR-T cells in peripheral blood using quantitative PCR and/or flow cytometry to assess expansion kinetics and persistence.
Serum cytokine profile | Baseline, Days 0-28, and at follow-up visits up to Month 12.
  Measurement of cytokine concentrations (e.g., IL-6, IFN-γ, TNF-α) in serum to monitor immune activation and correlate with clinical outcomes.

OTHER OUTCOMES:
Change in immune cell infiltration in tumor tissue (cells/mm²) | Baseline and approximately Day 28 post-infusion.
  Immune cell infiltration assessed in paired pre- and post-treatment tumor biopsies using multiplex immunofluorescence (MACSima platform). Cell density will be quantified as number of immune cells per mm² tumor tissue.
Microbiome diversity assessed by Shannon index | Baseline (pre-lymphodepletion) Day 0 (immediately before CAR-T infusion) Day 28 post-infusion
  Analysis of stool and tumor microbiome diversity using 16S rRNA sequencing and shotgun metagenomics. Microbiome diversity will be quantified using the Shannon diversity index.
Phenotype of innate-like T cell subsets in CAR-T products | At product release (Day 0) and follow-up samples up to Month 12.
  Characterization of γδ T cells, NKT cells, and MAIT cells in manufactured CAR-T products and their association with clinical outcome.
Change in CD318 antigen expression in tumor tissue (% positive tumor cells) | Baseline and approximately Day 28 post-infusion.
  CD318 expression assessed in paired pre- and post-treatment biopsies using spatial transcriptomics and proteomics. Reported as percentage of tumor cells expressing CD318.
Relative abundance of bacterial taxa in stool and tumor microbiome | Baseline (pre-lymphodepletion) Day 0 (before CAR-T infusion) Day 28 post-infusion
  Analysis of stool and tumor microbiome composition using 16S rRNA sequencing and shotgun metagenomics. Microbiome composition will be reported as the relative abundance (%) of bacterial taxa.

IPD SHARING:
Plan to Share IPD: No
At present, there are no plans to share individual participant data (IPD). Any potential future sharing of de-identified IPD will be considered in compliance with applicable laws and regulations, patient consent, and institutional policies. Should data sharing be implemented, information will be updated in this record accordingly.